CLINICAL TRIAL: NCT06728566
Title: Work at Heights Training: Conventional Approach With and Without Immersive Virtual Reality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Occidente (Other)
Collaborators: Universidad del Valle, Colombia (Other)
Responsible Party: Principal Investigator, Oscar Ivan Campo, Professor, Universidad Autonoma de Occidente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UAOccidente
Record Dates: First submitted 2024-10-24; First posted 2024-12-11 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Workers at Heights
Keywords: Occupational Groups; Virtual Reality; Simulation Training

STUDY DESIGN:
Intervention Model Description: The type of experimental design will be a Randomized Controlled Clinical Trial, with an analyst blind, to evaluate the efficacy and safety of the intervention. Participants will be randomly assigned to one of two groups, the group receiving the intervention, with work-at-heights training using immersive virtual reality, before practical training in a real field, and the control group, receiving the existing standard intervention (prior theoretical training only). This allows us to compare the results between the groups and determine if the intervention is effective compared to the control.
Who Masked: Outcomes Assessor
Masking Description: The analysts who perform the statistical analysis of the data will be blinded to the group assignments of the participants. This means that they will not know which participants received the immersive virtual reality training and which received the standard theoretical training. During data collection and management, the data will be anonymized and coded to prevent any identification of the participant's group assignment by those handling the data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inmersive virtual reality training (Experimental): Work at heights training with the addition of prior immersive virtual reality training.
  Interventions: Device: Inmersive virtual reality; Other: Conventional training
- Conventional training (Active Comparator): Training for work at heights using conventional strategy
  Interventions: Other: Conventional training

INTERVENTIONS:
Device: Inmersive virtual reality — In addition to conventional training, IVR training aims to provide a detailed preview of the tasks and procedures required in the standard training with selected virtual scenarios:
  Scenario 1: Inspection and Use of Personal Protective Equipment (PPE):
  In this scenario, the worker will inspect the equipment to ensure it is in good condition and properly used: Harness, Helmet, Lanyards, Carabiners, Lifelines, Energy Absorbers
  Scenario 2: Working on an Elevated Metal Structure:
  Structure Ascent: Ascent Method: Use specific ascent systems, ensuring you are always connected to an anchor point.
  Positioning on the Structure: Secure Anchorage: Once the working position is reached, secure the anchor to a fixed and reliable point.
  Structure Descent: Unanchoring and Reanchoring: Unanchor and re-anchor at secure points as you descend.
  Additional Safety Measures: Weather Conditions, signage and delimitation:
  Scenario 3: Rescue at Heights: Accessing the Person in Danger, rescue Techniques.
  Arms: Inmersive virtual reality training
Other: Conventional training — The working at heights training provided by the National Learning Service (SENA) in Colombia includes key steps to ensure safety and proper equipment use:
  * Harness Use: Inspect for damage, wear it like a vest, and ensure correct orientation. Adjust shoulder and leg straps for comfort and secure the chest strap.
  * Final Check: Verify D-rings are correctly positioned, and all buckles are securely fastened.
  * Helmet: Inspect for damage and adjust for a secure fit.
  * Lanyards: Select in good condition, connect properly, keep tension, and avoid overloading.
  * Carabiners: Use certified carabiners with functioning locks, connected to proper points.
  * Lifelines and Energy Absorbers: Install and tension lifelines properly; check energy absorbers before use.
  * Climbing/Descending: Maintain three contact points and secure tools to avoid accidents.

SUMMARY:
This study focuses on the design and evaluation of an innovative training protocol aimed at working at heights in the construction sector in the city of Cali. The main focus of this protocol lies in the use of Immersive Virtual Reality (IVR) and the measurement of biosignals to enhance workers' safety and preparedness. The training protocol is developed by creating virtual environments that simulate hazardous working conditions, allowing workers to practice high-risk situations safely and effectively. Additionally, the integration of biosignal measurements, such as heart rate variability and respiratory rate, is used to assess workers' stress levels and decision-making abilities during simulations.

The protocol evaluation is conducted through a pilot study with real workers in the construction field. The results are analyzed to determine whether the use of IVR and biosignal measurement improves assertiveness and, therefore, safety, reduces workplace accidents, and increases workers' confidence in high-risk environments. The findings of this study will provide valuable insights into the effectiveness of IVR and biosignal measurement as training tools in the construction sector, which could have a significant impact on reducing workplace accidents and injuries. This innovative approach has the potential to enhance occupational safety and workers' preparedness in high-risk environments, thereby contributing to a safer and more efficient working environment in the construction industry.

DETAILED DESCRIPTION:
Safety in the construction sector is of vital importance, especially in high-risk activities such as excavations and working at heights. To improve worker training and preparation in these areas, this research proposal has been developed.

This project focuses on the use of advanced technology, such as Immersive Virtual Reality, to simulate real work situations and allow workers to practice and acquire the necessary skills to face the challenges of their daily tasks. However, what makes this project particularly interesting is the incorporation of biosignal measurement during training.

Biosignals are physiological indicators that can be measured and analyzed to assess an individual's emotional and physical state. In this context, devices will be used to capture data such as heart rate, respiratory rate, and their variability. These measurements will provide precise information about the worker's reactions to different simulated situations, which will, in turn, help identify areas for improvement and optimize the training protocol.

The main contribution of this project lies in generating new knowledge about how biosignals can be used as a complementary tool in the design and evaluation of training protocols for workers in high-risk activities. The information obtained through biosignal measurement will allow for the identification of patterns and trends that will help better understand workers' physiological and emotional reactions, as well as their performance in critical situations.

This clinical trial compares two training methods for workers at heights, one using Immersive Virtual Reality (IVR) in addition to the conventional training, and the other using only the conventional training. The main questions to be answered are:

What is the impact of the IVR training protocol on the acquisition of knowledge and practical skills of workers in high-risk activities compared to traditional training?

Is there a relationship between immersive Virtual Reality training and the physiological response to stressful situations in high-risk activities, through the recording of biosignals taken during the intervention?

The researchers will compare the two forms of training and identify if there are differences in both fitness and cardiorespiratory response.

Participants in the control group will perform practical work at heights while heart rate, respiratory monitoring, and ergonomic analysis of the activity will be performed. The participants of the intervention group, in addition to the above, will be exposed to virtual reality environments as part of the training of work at heights, this will be before the actual practical part.

ELIGIBILITY:
Inclusion Criteria:

* Learners from the National Learning Service (SENA).
* First time taking the work at heights training course.

Exclusion Criteria:

* Experience in working at heights.
* Health conditions that prevent performing both the IVR training and work at heights.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
PRACTICAL SKILLS FOR WORKING AT HEIGHTS | The time frame for completing all practical activities, assessments, and evaluations is approximately 10 hours, distributed over 2 days.
  Each activity is scored on an approve/disapprove system. By the end, workers must meet these standards:
  1. Harness Donning and Adjustment: Properly don, adjust straps, and ensure no slack. Passing requires a secure, comfortable fit and correct anchor positioning.
  2. Anchor Points: Select/install anchors compatible with the system and load standards. Passing requires secure installation verified by testing.
  3. Lifelines: Use vertical/horizontal lifelines, maintaining connection. Passing requires constant security.
  4. Climbing/Moving: Safely ascend/descend while connected. Passing requires proper system use and controlled movements.
  5. Tool Handling: Secure tools to prevent falls. Passing requires consistent adherence to safety protocols.
  6. Emergency Response: Simulate emergencies calmly, following protocols. Passing requires appropriate stress management.
  7. Equipment Inspection: Identify equipment issues. Passing requires thorough inspection and defect reporting.

SECONDARY OUTCOMES:
Heart Rate Variability | Heart rate variability will be assessed over an approximate period of 45 minutes.
  Variation in the time between RR intervals on the electrocardiogram
Respiratory Rate Variability | Respiratory rate variability will be assessed over an approximate period of 45 minutes.
  The fluctuation in time between consecutive breathing cycles.
Ergonomic Analysis of the Activity | The REBA score will be assessed over an approximate period of 25 minutes during the observation of the occupational task.
  The REBA (Rapid Entire Body Assessment) score quantifies the ergonomic risk of musculoskeletal injury in occupational tasks by evaluating body postures, forces, and repetitive movements. It assigns values to the position of the head, torso, arms, legs, and wrists, physical effort (e.g., lifting, pushing, pulling), and task repetition. The total score ranges from 1 to 15, with scores from 1-3 indicating minimal risk, 4-7 indicating moderate risk, and 8-15 suggesting high risk. A higher REBA score indicates greater potential for musculoskeletal disorders. The REBA score helps identify ergonomic risks and prioritize interventions to reduce injury risk.
Attention and memory measurements | Before the training protocol
  The Neuropsi (Neuropsychological Screening Battery) score assesses cognitive function in multiple domains, including attention, memory, executive function, and language. It consists of tasks measuring short-term memory, attention span, visuospatial abilities, and verbal fluency, among others. The total score is calculated by summing the results from each subtest, with a range from 0 to 30 points for each domain. Higher scores indicate better cognitive performance, while lower scores suggest cognitive impairment. The Neuropsi score is used to monitor cognitive changes over time and evaluate the effectiveness of therapeutic interventions. A score below 20 typically indicates significant cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Campo, PhD, Study Director — Universidad Autónoma de Occidente

IPD SHARING:
Plan to Share IPD: Yes
Once the research is completed, only data that are useful for obtaining results will be stored in www.figshare.com and placed under embargo until they are published in a scientific journal. No sensitive or personal data will be uploaded to this repository.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be open access once it has been approved for publication in a scientific journal, these data will be permanently available.
Access Criteria: The data will be open access, only information relevant to the research objectives will be included. No identifying data or any other sensitive data will be included.
URL: http://www.figshare.com

REFERENCES:
- [Background] Abrahamsen EB, Selvik JT, Milazzo MF, Langdalen H, Dahl RE, Bansal S, et al. On the use of the 'Return Of Safety Investments' (ROSI) measure for decision-making in the chemical processing industry. Reliab Eng Syst Saf. 2021 Jun 1;210:107537.
- [Background] Nnaji C, Okpala I, Gambatese J, Jin Z. Controlling safety and health challenges intrinsic in exoskeleton use in construction. Saf Sci. 2023 Jan 1;157:105943.
- [Background] Bao L, Tran SVT, Nguyen TL, Pham HC, Lee D, Park C. Cross-platform virtual reality for real-time construction safety training using immersive web and industry foundation classes. Autom Constr. 2022 Nov 1;143:104565.
- [Background] Zermane A, Mohd Tohir MZ, Baharudin MR, Mohamed Yusoff H. Risk assessment of fatal accidents due to work at heights activities using fault tree analysis: Case study in Malaysia. Saf Sci. 2022 Jul 1;151:105724.
- [Background] Stefan H, Mortimer M, Horan B, Kenny G. Evaluating the preliminary effectiveness of industrial virtual reality safety training for ozone generator isolation procedure. Saf Sci. 2023 Jul 1;163:106125.
- [Background] Shakerian S, Habibnezhad M, Ojha A, Lee G, Liu Y, Jebelli H, et al. Assessing occupational risk of heat stress at construction: A worker-centric wearable sensor-based approach. Saf Sci. 2021 Oct 1;142:105395.

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT06728566/SAP_000.pdf
  • Informed Consent Form (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/66/NCT06728566/ICF_001.pdf